CLINICAL TRIAL: NCT02292511
Title: Mind-motor Exercise in Older Adults With Type 2 Diabetes and Self-reported Cognitive Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Rob Petrella, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D-SSE-123
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: subjective cognitive impairment; mind-motor intervention; square-stepping exercise; older adults
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Square-Stepping Exercise Intervention (Experimental): Participants in this group will attend a square-stepping exercise intervention 60 minutes on two days a week at a community location.
  Interventions: Behavioral: Square-stepping exercise
- Usual-care wait-list control (No Intervention): This group will receive standard care and be invited to partake in the intervention after all assessments have been completed.

INTERVENTIONS:
Behavioral: Square-stepping exercise — In a group setting, an instructor will demonstrate walking patterns on a gridded mat to the participants and the participants must memorize and repeat the patterns on their own. This program has over 200 patterns that increase in difficulty from beginner to advanced. Eighty percent of the group must successfully complete the patterns to move onto the next pattern. Social engagement is encouraged.
  Other Names: mind-motor exercise
  Arms: Square-Stepping Exercise Intervention

SUMMARY:
The purpose of this study is to determine if a 6 month mind-motor intervention will help to improve overall brain health in adults over the age of 55 with type 2 diabetes and a self-reported complaint about memory or thinking skills. It is hypothesized that the intervention group will show improvements in their overall brain health after 6 months of mind-motor training compared to the control group.

DETAILED DESCRIPTION:
Dementia has been identified as a global health concern because of the increase in incidence globally. Regardless of whether individuals with self-reported cognitive complaints (CCs) have objective impairment, they are at increased risk for cognitive decline, and they are comparable to those with early mild cognitive impairment (MCI) for brain atrophy and increased risk of progression towards Alzheimer's disease (AD). People who express being worried about their memory or cognition show a further increased risk of cognitive decline. If prevention programs could delay the onset of dementia even in part of the at-risk population, this could decrease disease prevalence significantly. The risk of cognitive impairment or dementia is increased in type 2 diabetes (T2D) and T2D accelerates the progression from MCI to dementia.

The proposed mind-motor intervention for the prevention of cognitive decline in T2D is called square stepping exercise (SSE). The SSE program was developed by Shigematsu and Okura (2005) and can be best described as a visuospatial working memory task with a stepping response. There are more than 200 patterns developed for this program that progress from simple to advanced stepping patterns. The primary focus of Shigematsu and colleagues' research has been to examine the impact of SSE on fall risk factors and mobility in older adults. Within their research they have found that SSE improves lower extremity functional fitness, reduces fall risk, and improves overall fitness in older adults when compared to walking or strength and balance training. In combination with Dr. Shigematsu's research in Japan in healthy older adults, the investigators are aiming to provide a significant evidence base for SSE internationally and within varied populations, including older adults with subjective cognitive complaints and with different chronic diseases. In collaboration with Dr. Shigematsu, the investigators have executed SSE studies at the Canadian Centre for Activity and Aging and currently are running a study in the community in Woodstock, ON. Preliminary evidence has shown that over a 6-month exercise plus mind-motor training period, participants improved in global cognitive functioning, verbal learning and memory, and verbal fluency, when compared to an exercise control group. Most recently, Shigematsu and colleagues have found the SSE program to improve memory and executive function in a 6-month pilot study.

The overarching goal of the investigators is healthy aging; research goals aim to evaluate intervention tools in the prevention of cognitive decline at one of the earliest markers of cognitive decline, which is a subjective complaint. As well, goals of the intervention strategies are to maintain mobility and balance with advancing age and chronic disease. The T2D population is at increased risk of decline and the added component of self-management of diabetes and insulin treatment makes it crucial to maintain adequate cognition and independence in this population.

Study Design: This study will be a 24-week Proof-of-Concept randomized controlled trial (1:1 allocation) whereby consenting and eligible participants will be randomized to either: 1) the SSE intervention group or 2) a usual-care, wait-list control group. Participants will be recruited from the St. Joseph's Primary Care Diabetes Support Program (SJHC- PCDSP) and the study intervention will be conducted at a community location in London, Ontario. This will be a single blinded study. All assessments will be done pre-intervention (V0) and post-intervention (V2), with interim assessments after 12-weeks (V1) (with the exception of sensorimotor). Assessments will take place at SJHC-PCDSP and Western University. One assessment will be done online either at the participant's home or at SJHC-PCDSP (solely completed by the participant)(i.e. Cambridge Brain Sciences). We will use blocked randomization and thus, participants will begin and complete the trial within waves.

Participants: All participants will be required to self-report a cognitive complaint; once eligibility is determined, participants will then be asked further questions about their cognition. Participants will undergo a number of measurements at baseline, which will be used to describe the study sample. These measures include: i) baseline cognition: Montreal Cognitive Assessment (MoCA) and the Clock Drawing Test; ii) baseline fitness: Step test iii) Anthropometric measures: weight, height, waist circumference; iv) history of physical and mental activities: Leisure Activities questionnaire v) clinic blood work values HbA1c, creatine (eGFR), and lipid assessment obtained from clinic electronic medical records (EMR) and vi) demographic information. Current medications, blood pressure and patient medical history will also be obtained from EMRs.

Intervention SSE (Intervention) Group: Participants in the Square Stepping Exercise group will be doing a group-based mind-motor intervention program. Participants will come to a community location for 60 minutes on one day per week to participate in the SSE program. An instructor will be present to demonstrate the walking patterns on a gridded mat. Participants must memorize and complete the patterns as a group, and they are encouraged to help one another to promote social engagement. Eighty percent of the group must successfully complete the patterns to move on to the next pattern. There are over 200 patterns that increase in difficulty from beginner, to intermediate and advanced. If some participants are struggling to keep up with the group, a catch-up session will be made available to assist those participants. Participants will be asked to use the smartphone application (Healthebrain) 10 minutes per day or 2 patterns as homework to supplement the SSE program. Participants will be able to use their own smartphones (apple or android devices) or they will be given a smartphone to use for the duration of the study as needed.

Wait-List Control Group: The investigators have opted to use a wait-list control group for this study in order to see differences of our intervention from usual care in T2D.The control group will be on a wait list to participate in the 24-week SSE program, which will commence after all measurements are completed by both groups. The classes will be offered free of charge.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years of age or older
* Stable type 2 diabetes (i.e. A1c <9.0 for at least 6 months)
* Self report a cognitive complaint (i.e answer yes to: do you feel your memory and/or thinking skills have gotten worse recently?)

Exclusion Criteria:

Participants must be able to comprehend the letter of information and provide consent.

Participants cannot have

* major depression, measured by Center of Epidemiologic Studies Depression Scale (CES-D) and study physician consult,
* diagnosis of dementia, or score <24 on mini-mental state examination (MMSE)
* other significant neurological disorder or psychiatric conditions
* severe history of cardiovascular events
* severe orthopedic limitations
* uncontrolled diabetes (i.e A1c <4.0mmol/L or >9.0mmol/L)
* unstable angina
* untreated retinopathy
* foot ulcers with or without severe peripheral neuropathy
* severe sensory impairment (i.e. blind).

Finally, participants must plan to attend at least 75% of the sessions over the 24-week period; this is to ensure adequate compliance of the program.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Global Cognitive Functioning | Change from 0 to 24 weeks
  measured by Cambridge Brain Sciences - composite score from 12 tasks

SECONDARY OUTCOMES:
Global Cognitive Functioning | Change from 0 to 12 weeks
  measured by Cambridge Brain Sciences - composite score from 12 tasks
Memory composite score | Change from 0 to 12 & 24 weeks
  measured by Cambridge Brain Sciences - composite score from 4 memory tasks
Reasoning composite score | Change from 0 to 12 & 24 weeks
  measured by Cambridge Brain Sciences - composite score from 3 reasoning tasks
Concentration composite score | Change from 0 to 12 & 24 weeks
  measured by Cambridge Brain Sciences - composite score from 3 concentration tasks
Planning (executive functioning) composite score | Change from 0 to 12 & 24 weeks
  measured by Cambridge Brain Sciences - composite score from 2 planning (executive function) tasks
Gait Speed | Change from 0 to 12 & 24 weeks
  measured by 6 metre walk test
Prosaccade reaction time | Change from 0 to 24 weeks
  measured by eye tracking - the reaction time of the eye when instructed to look toward a flash of light
Antisaccade reaction time | Change from 0 to 24 weeks
  measured by eye tracking - the reaction time of the eye when instructed to look away from a flash of light
Prosaccade direction errors | Change from 0 to 24 weeks
  measured by eye-tracking - the amount of eye movement error on trials
Antisaccade direction errors | Change from 0 to 24 weeks
  measured by eye-tracking - the amount of eye movement error on trials

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Petrella, MD, PhD, Principal Investigator — University of Western Ontario, Lawson Health Research Institute
Locations (1):
- St. Joseph's Primary Care Diabetes Support Program, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No